CLINICAL TRIAL: NCT03834948
Title: A Phase 1/2 Multicenter, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of AO-176
Brief Title: AO-176 in Multiple Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arch Oncology (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AO-176-101; KEYNOTE-C49 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor
Keywords: CD47; AO-176; Immunotherapy
MeSH Terms: interventions — Paclitaxel; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Each dose escalation cohort will initially recruit 3 patients to receive AO-176 or AO-176 + paclitaxel or AO-176 + pembrolizumab in a standard 3+3 design; the cohort will be expanded in the event of a DLT.
  Once the MTD/RP2D has been established for monotherapy, AO-176 + paclitaxel or AO-176 + pembrolizumab, tumor-specific dose expansion cohorts will be recruited to further assess safety and evaluate preliminary efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- AO-176 Dose Escalation (Experimental): Each dose escalation cohort will initially recruit 3 patients to receive AO-176 in a standard 3+3 design; cohorts will be expanded in the event of a DLT.
  Interventions: Drug: AO-176
- AO-176 Dose Expansion (Experimental): Once the MTD/RP2D has been established, tumor-specific dose expansion cohorts will be recruited to further assess safety and evaluate preliminary efficacy of AO-176.
  Interventions: Drug: AO-176
- AO-176 + Paclitaxel Dose Escalation (Experimental): Each dose escalation cohort will initially recruit 3 patients to receive AO-176 and paclitaxel in a standard 3+3 design; cohorts will be expanded in the event of a DLT.
  Interventions: Drug: AO-176 + Paclitaxel
- AO-176 + Paclitaxel Dose Expansion (Experimental): Once the MTD/RP2D has been established, tumor-speciﬁc dose expansion cohorts will be recruited to further assess safety and evaluate preliminary efﬁcacy of AO-176 + paclitaxel.
  Interventions: Drug: AO-176 + Paclitaxel
- AO-176 + Pembrolizumab Dose Escalation (Experimental): Each dose escalation cohort will initially recruit 3 patients to receive AO-176 and pembrolizumab in a standard 3+3 design; cohorts will be expanded in the event of a DLT.
  Interventions: Drug: AO-176 + Pembrolizumab
- AO-176 + Pembrolizumab Dose Expansion (Experimental): Once the MTD/RP2D has been established, tumor-speciﬁc dose expansion cohorts will be recruited to further assess safety and evaluate preliminary efﬁcacy of AO-176 + pembrolizumab.
  Interventions: Drug: AO-176 + Pembrolizumab

INTERVENTIONS:
Drug: AO-176 — Humanized monoclonal antibody (mAb) targeting CD47
  Arms: AO-176 Dose Escalation; AO-176 Dose Expansion
Drug: AO-176 + Paclitaxel — Humanized monoclonal antibody (mAb) targeting CD47 and paclitaxel
  Arms: AO-176 + Paclitaxel Dose Escalation; AO-176 + Paclitaxel Dose Expansion
Drug: AO-176 + Pembrolizumab — Humanized monoclonal antibody (mAb) targeting CD47 and pembrolizumab
  Arms: AO-176 + Pembrolizumab Dose Escalation; AO-176 + Pembrolizumab Dose Expansion

SUMMARY:
This is a first-in-human, Phase 1/2 multi-center, open-label, dose escalation and expansion study of AO-176 which will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and clinical effects of AO-176 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1/2 multicenter, open-label, dose escalation and expansion study of AO-176 in patients with solid tumors. Part A of this study will examine escalating repeat doses of AO-176 monotherapy in patients with select advanced solid tumors, including epithelial ovarian carcinoma (EOC), which will include primary peritoneal and fallopian tube carcinoma; squamous cell carcinoma of the head and neck; endometrial carcinoma; castration resistant prostate cancer; non-small cell lung adenocarcinoma; papillary thyroid carcinoma; pleural or peritoneal malignant mesothelioma; and gastroesophageal adenocarcinoma, for which standard therapy proven to provide clinical benefit does not exist or is no longer effective.

Part B and Part C of this study will examine escalating repeat doses of AO-176 in combination with paclitaxel (Part B) or pembrolizumab (Part C) in platinum-resistant EOC, including primary peritoneal and fallopian tube carcinoma; endometrial carcinoma; and gastric adenocarcinoma/gastroesophageal adenocarcinoma.

The monotherapy and combination dose escalation portions of the study utilize a classic 3+3 design, with enrollment of 3 patients per cohort and expansion of the cohort in the event of a dose-limiting toxicity (DLT).

Once the maximum-tolerated dose (MTD)/recommended phase 2 dose (RP2D) has been established in dose escalation, tumor-specific dose expansion cohorts will be recruited to further assess safety and evaluate preliminary efficacy of AO-176 as monotherapy, in combination with paclitaxel, and in combination with pembrolizumab.

ELIGIBILITY:
Key Inclusion Criteria

1. Select advanced solid tumor for which standard therapy proven to provide clinical benefit does not exist, or is no longer effective

   Part A:
   * Epithelial ovarian carcinoma (EOC)
   * Endometrial carcinoma
   * Castration resistant prostate cancer
   * Non-small cell lung adenocarcinoma
   * Papillary thyroid carcinoma
   * Malignant mesothelioma (pleural or peritoneal)
   * Gastroesophageal adenocarcinoma
   * Squamous cell carcinoma of the head and neck

   Part B and Part C:
   * Platinum-resistant EOC (including fallopian tube or primary peritoneal cancer)
   * Endometrial carcinoma
   * Gastric adenocarcinoma/gastroesophageal adenocarcinoma
2. Measurable disease
3. ECOG status 0-1
4. Resolution of prior-therapy-related adverse effects
5. Minimum of 4 weeks or 5 half-lives since last dose of cancer therapy

Key Exclusion Criteria:

1. Previous hypersensitivity reaction to treatment with another monoclonal antibody
2. Unresolved hypersensitivity to paclitaxel or any of its excipients (Part B only). Patients who have been desensitized may participate.
3. Part C Only

   1. History of interstitial lung disease or a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
   2. History of immune mediated colitis, hepatitis, endocrinopathies, nephritis or significant immune mediated skin reactions such as toxic epidermal necrolitis or Stevens -Johnson Syndrome
   3. History of any autoimmune disease which required systemic therapy* in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs) including but not limited to: i. Inflammatory bowel disease (including ulcerative colitis and Crohn's Disease) ii. Rheumatoid arthritis iii. Systemic progressive sclerosis (scleroderma) iv. Systemic lupus erythematosus v. Autoimmune vasculitis (e.g. Wegener's granulomatosis) *Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed)
4. Prior treatment with a checkpoint inhibitor (anti-PD-1, PD-L1, CTLA-4 etc.) within 4 weeks prior to the start of study drug
5. Prior treatment with a CD47-targeted therapy
6. Prior organ or stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Safety of AO-176 assessed by adverse events and laboratory abnormalities | Up to 12 months
  Evaluate the safety of AO-176 measured by the number adverse events, serious adverse events and lab abnormalities.
Safety of AO-176 and paclitaxel assessed by adverse events and laboratory abnormalities | Up to 12 months
  Evaluate the safety of AO-176 in combination with paclitaxel measured by the number adverse events, serious adverse events and lab abnormalities.
Safety of AO-176 and pembrolizumab assessed by adverse events and laboratory abnormalities | Up to 12 months
  Evaluate the safety of AO-176 in combination with pembrolizumab measured by the number adverse events, serious adverse events and lab abnormalities.

SECONDARY OUTCOMES:
AO-176 anti-tumor activity assessed by changes in response criteria | Up to 12 months
  Evaluate objective response rate of AO-176 using RECIST v1.1 and iRECIST.
AO-176 + paclitaxel anti-tumor activity assessed by changes in response criteria | Up to 12 months
  Evaluate objective response rate of AO-176 in combination with paclitaxel using RECIST v1.1 and iRECIST.
AO-176 + pembrolizumab anti-tumor activity assessed by changes in response criteria | Up to 12 months
  Evaluate objective response rate of AO-176 in combination with pembrolizumab using RECIST v1.1 and iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Benajmin Oshrine, MD, Study Director — Arch Oncology
Locations (10):
- United States (10):
  - University of Southern California, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Oklahoma University, Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health Science University, Portland, Oregon
  - Sidney Kimmel Cancer Center, Thomas Jefferson University, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Northwest Medical Specialties, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andrejeva G, Capoccia BJ, Hiebsch RR, Donio MJ, Darwech IM, Puro RJ, Pereira DS. Novel SIRPalpha Antibodies That Induce Single-Agent Phagocytosis of Tumor Cells while Preserving T Cells. J Immunol. 2021 Feb 15;206(4):712-721. doi: 10.4049/jimmunol.2001019. Epub 2021 Jan 11. PMID 33431660